CLINICAL TRIAL: NCT07197853
Title: A Prospective, Single-Center, Randomized Controlled Trial to Evaluate the Clinical Efficacy and Safety of Microwave Ablation Combined With Huaier Granules in Patients With Stage IA Non-Small Cell Lung Cancer
Brief Title: Clinical Efficacy and Safety of Microwave Ablation Combined With Huaier Granules in Patients With Inoperable Stage IA Non-Small Cell Lung Cancer: A Prospective, Single-Center, Randomized Controlled Clinical Trial
Acronym: HAMSTER
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xin Ye (Other)
Responsible Party: Sponsor-Investigator, Xin Ye, professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HAMSTER
Record Dates: First submitted 2025-09-26; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Non-small Cell Lung Cancer (NSCLC); Huaier Granules; Microwave Ablation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MWA + huaier (Experimental): MWA + huaier
  Interventions: Drug: Huaier Granule
- MWA (Experimental): MWA
  Interventions: Drug: Huaier Granule

INTERVENTIONS:
Drug: Huaier Granule — Patients in this arm will undergo CT-guided percutaneous microwave ablation using a standard protocol (2450 MHz, 30-50 W, 5-10 minutes per lesion, multi-probe as needed based on tumor size). Seven days post-ablation, patients will start oral administration of Huaier granules at a dose of 10g, three times daily (TID), for 72 consecutive weeks. The combined therapy aims to improve local tumor control and modulate anti-tumor immunity.

SUMMARY:
This prospective, single-center, randomized controlled clinical trial aims to evaluate the efficacy and safety of microwave ablation (MWA) combined with Huaier granules in patients with inoperable stage IA non-small cell lung cancer (NSCLC). A total of 180 eligible patients will be randomly assigned to receive either MWA alone or MWA combined with Huaier granules. The primary endpoint is progression-free survival (PFS) assessed by RECIST 1.1 criteria. Secondary outcomes include local progression rate (LPR), overall survival (OS), tumor markers, immune function, and quality of life. Safety will be evaluated using the CTCAE v5.0 criteria. The study seeks to determine whether the combined therapy offers improved tumor control and immune benefits over MWA alone.

DETAILED DESCRIPTION:
Lung cancer remains the leading cause of cancer-related death globally, with non-small cell lung cancer (NSCLC) accounting for approximately 85% of cases. A significant proportion of early-stage NSCLC patients are deemed inoperable due to comorbidities or patient refusal. Microwave ablation (MWA) is an established local therapy for inoperable NSCLC, yet incomplete ablation and immune suppression in the tumor microenvironment remain challenges, especially in tumors >3 cm or near critical structures.

This study investigates whether the addition of Huaier granules, a polysaccharide-based traditional Chinese medicine shown to modulate immune function and improve outcomes post-ablation in liver cancer, can enhance the efficacy of MWA in early-stage NSCLC. Huaier may promote dendritic cell maturation, Th1 immune responses, and restore immune balance after incomplete MWA (iMWA).

Eligible patients (stage IA-IIA NSCLC without lymph node metastasis, ECOG ≤2, life expectancy >3 months) will be randomized 1:1 into two groups. The experimental group will receive CT-guided MWA followed by oral Huaier granules (10 g three times daily for 72 weeks), while the control group receives MWA alone. Follow-up will occur at months 1, 3, 6, 12, and 24.

Primary endpoint: progression-free survival (PFS). Secondary endpoints: local progression rate (LPR), overall survival (OS), immune cell profiles, tumor markers (e.g., CEA, CYFRA21-1), and quality of life (EORTC QLQ-C30/LC13).

Safety will be monitored via laboratory tests and adverse event reporting according to CTCAE v5.0.

The trial is expected to provide high-level evidence on whether the integration of Huaier granules into MWA-based therapy improves clinical outcomes and immune recovery in early inoperable NSCLC.

ELIGIBILITY:
Inclusion Criteria

Age:

≥ 18 years old.

Diagnosis:

Histologically or cytologically confirmed IA stage non-small cell lung cancer (NSCLC) that is inoperable.

ECOG Performance Status:

0-2 (Eastern Cooperative Oncology Group performance status).

Previous Treatment:

Patients must have received no prior systemic treatment for lung cancer.

Informed Consent:

Ability to provide written informed consent and willingness to comply with study requirements.

Adequate Organ Function:

Patients must have adequate hepatic, renal, and hematologic function as evidenced by:

Bilirubin ≤ 1.5 × upper limit of normal (ULN)

ALT/AST ≤ 2.5 × ULN

Creatinine clearance ≥ 30 mL/min

Absolute neutrophil count (ANC) ≥ 1,500 cells/μL

Exclusion Criteria

Other Malignancies:

Active or history of other malignancies within the past 5 years, except for non-melanoma skin cancer or in situ carcinoma.

Severe Concurrent Diseases:

Any serious or uncontrolled medical condition such as:

Cardiovascular disease (e.g., recent myocardial infarction, unstable angina, or severe arrhythmia)

Uncontrolled diabetes or hypertension

Active infections requiring systemic antibiotics or antivirals

Pregnancy or Breastfeeding:

Women who are pregnant, breastfeeding, or planning to become pregnant during the study.

Immunosuppressive Therapy:

Patients who have received immunosuppressive therapy within 30 days prior to enrollment.

Other Contraindications:

Known hypersensitivity to any of the components of the treatment regimen (e.g., microwave ablation, Huai Er Granules).

Other Unspecified Conditions:

Any other condition or circumstances that, in the investigator's opinion, may interfere with the study or pose a risk to the patient.

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 24 months after treatment initiation
  PFS is defined as the time from randomization to disease progression or death from any cause, whichever occurs first. Disease progression will be assessed based on RECIST 1.1 criteria through imaging evaluations. Patients who are alive and progression-free at the time of analysis will be censored at their last disease assessment.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol